CLINICAL TRIAL: NCT06590116
Title: Patient and Physical Therapist Perspectives on Spinal Manipulative Therapy for Low Back Pain
Brief Title: Perspectives on Spinal Manipulative Therapy for Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202301700
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Patients seeking physical therapy for low back pain
  Interventions: Other: Physical therapy
- Physical therapists (Other): Physical therapists treating enrolled patients
  Interventions: Other: Physical therapist provider

INTERVENTIONS:
Other: Physical therapy — Patients with low back pain will receive a combination of education, spinal manipulative therapy, and exercise as prescribed by their physical therapist
  Arms: Patients
Other: Physical therapist provider — Physical therapists will provide a combination of education, spinal manipulative therapy, and exercise to their patients with low back pain participating in the study
  Arms: Physical therapists

SUMMARY:
The goal of this study is to better understand how the thoughts and beliefs of patients with low back pain and their physical therapist influence how much patients benefit from physical therapy. Participants will receive physical therapy as determined by their physical therapist including spinal manipulative therapy, exercise, and education. Participants with low back pain and their physical therapists will complete forms about their thoughts and beliefs about low back pain and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pain between 12th rib and buttocks with or without symptoms into one or both legs, which, in the opinion of the examiner, originate from the lumbar region.
* Meets NIH Task Force criteria for chronic low back pain

Exclusion Criteria:

* Prior surgery to the lumbosacral spine
* Currently pregnant
* Not currently receiving spinal manipulative therapy or exercise interventions from another healthcare provider such as a chiropractor or massage therapist.
* No neurogenic signs indicating radiculopathy
* No "red flags" of a potentially serious condition (e.g., cauda equina syndrome, fracture, cancer, infection, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
PROMIS-29 | Baseline and 2 weeks and 6 weeks and 12 weeks and 18 weeks and 26 weeks
  Assesses pain intensity using a single item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. This will only be completed by patient participants in the study.
NIH Chronic LBP Impact Score | 12 weeks and 26 weeks
  Combines results of the Pain Intensity, Physical Function, and Pain Interference PROMIS scores. Scores range from 8 (least impact) to 50 (greatest impact).

SECONDARY OUTCOMES:
Patient Acceptable Symptom State | Baseline and 2 weeks and 6 weeks and 12 weeks and 18 weeks and 26 weeks
  The PASS is a self-report, single item question asking: "Taking into account the many ways your pain affects your daily life, if you were to remain for the next few months as you are now, would you consider your current state to be satisfactory?" with response options being 'Yes' or 'No'. Only patient participants will complete this assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Beneciuk JM, Bialosky J, Hayes JR, Buzzanca-Fried KE, Rowe R, Cristello S, Harrison T, Vickers R, Shan G. Patient and physical therapist perspectives on spinal manipulative therapy for low back pain and associated clinical outcomes: protocol for a prospective, single-arm intervention study. BMJ Open. 2025 Jul 11;15(7):e099932. doi: 10.1136/bmjopen-2025-099932. PMID 40645636